CLINICAL TRIAL: NCT05501860
Title: A Randomized, Double-Masked, Placebo-Controlled, Parallel-Group Evaluation of the Ocular Safety of Articaine Sterile Topical Ophthalmic Solution
Brief Title: A Safety Study of of AG-920 Sterile Topical Ophthalmic Solution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Genomics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AG-920-CS303
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia, Local
Keywords: AG-920; Articaine; Septocaine
MeSH Terms: interventions — Carticaine

STUDY DESIGN:
Intervention Model Description: Subjects who provide informed consent and fulfill all the inclusion criteria and none of the exclusion criteria will be randomized in a 2:1 ratio to receive a single dose of AG-920 or placebo into one (study) eye (2 drops 30 seconds apart).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study is double masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AG-920 (Experimental): Articaine Sterile Topical Ophthalmic Solution (AG-920) is a sterile, isotonic, non-preserved aqueous solution containing the active ingredient Articaine HCl 8%.
  Interventions: Drug: AG-920
- Placebo (Placebo Comparator): Placebo Sterile Topical Ophthalmic Solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AG-920 — AG-920 Sterile Topical Ophthalmic Solution
  Other Names: articaine
  Arms: AG-920
Drug: Placebo — Placebo Sterile Topical Ophthalmic Solution
  Arms: Placebo

SUMMARY:
A Phase 3, randomized, placebo-controlled, double-masked, parallel study in healthy subjects. It is designed to evaluate the ocular safety of a single topical ocular administration of AG-920 sterile topical ophthalmic solution compared to placebo..

DETAILED DESCRIPTION:
A Phase 3, randomized, placebo-controlled, double-masked, parallel study in healthy subjects performed in the US. It is designed to evaluate the ocular safety of one dose of AG-920 compared to placebo. I). In this study, subjects who provide informed consent and fulfill all the inclusion criteria and none of the exclusion criteria will be randomized in a 2:1 ratio to receive one dose of AG-920 or identical looking placebo into one (study) eye. A subset of subjects will undergo endothelial cell count (ECC) evaluations.

Each dose of AG-920 or placebo will consist of two drops in the study eye. After the completion of dosing, subjects will undergo a series of eye exams that will be documented. Investigational medicinal product (IMP) dosing will be performed by the study staff.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study-related procedures being performed.
2. Male or a non-pregnant, non-lactating female.
3. Healthy by clinical assessment, including ocular examination.
4. Have an Early Treatment of Diabetic Retinopathy Study (ETDRS) best corrected visual acuity (BCVA) of 20/200 or better in both eyes.
5. Have an Intraocular Pressure (IOP) between 7 and 30 mmHg.

   Specular microscopy subset subjects only:
6. Have a central corneal endothelial cell density of ≥1500 cells/mm2 at baseline

Exclusion Criteria:

1. . Have participated in an investigational study within the past 30 days.
2. Have a contraindication to local anesthetics, Septocaine®, or any component of the IMP.
3. Have had ocular surgery or general surgery in either eye within the past 90 days.
4. Have had an intravitreal injection in either eye within 14 days of randomization.
5. Have ocular surface disease requiring punctal plugs.
6. Have evidence of any current ocular inflammation.
7. Current ocular allergy symptoms.
8. Have used topical, ocular medications in the 24 hours preceding dosing.
9. Systemic opioid, opiate analgesic or topical Non-steroidal Anti-Inflammatory Drug (NSAID) use within the past 30 days.
10. Previous participation in a clinical study of AG-920.
11. A current condition which could cause vision problems such as Pseudotumor Cerebri.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Uram, MD, Study Director — Medical Expert
Locations (2):
- United States (2):
  - American Genomics Site 1, Newport Beach, California
  - American Genomics Site 2, McAllen, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Studied Period: 30 July 2022 to 7 December 2022 @ two study centers in the US.
Period: Overall Study
Arm/Group | AG-920 | Placebo
Started | 166 | 83
Specular Microscopy Population | 13 | 3
Completed | 165 | 82
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AG-920 | Placebo | Total
Number analyzed (Participants) | 166 | 83 | 249
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 149 | 74 | 223
  >=65 years | 17 | 9 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (16.3) | 40.1 (15.8) | 39.6 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 48 | 154
  Male | 60 | 35 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 118 | 56 | 174
  Not Hispanic or Latino | 48 | 27 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 13 | 5 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 153 | 75 | 228
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 166 | 83 | 249
Study Eye [Count of Participants; unit: Participants]
  Left Eye (OS) | 83 | 42 | 125
  Right Eye (OD) | 83 | 41 | 124
Color of Iris [Count of Participants; unit: Participants]
  Blue | 11 | 7 | 18
  Brown | 128 | 66 | 194
  Green | 13 | 3 | 16
  Hazel | 14 | 7 | 21
BCVA LogMar [Mean (Standard Deviation); unit: LogMar]
  BCVA LogMar Study Eye | 0.0 (0.2) | 0.0 (0.2) | 0.0 (0.2)
  BCVA LogMar Fellow Eye | 0.0 (0.2) | 0.0 (0.2) | 0.0 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs will be summarized by treatment group using frequency and percent for each system, organ, class (SOC) and preferred term within each SOC.
Time Frame: From Day 1 (treatment day) to 4 days following treatment day; 90 days following treatment for subjects participating in specular microscopy.
Population: The safety population is defined as all subjects which were randomized and who received at least one drop of the dose (2 drops) of the study medication. The ITT population is defined as all subjects who were randomized to treatment and have received at least one dose (two drops) of the study medication. In this study, the ITT and safety populations were found to be identical.
Measure: Count of Participants; unit: Participants
Arm/Group | AG-920 | Placebo
Number analyzed (Participants) | 166 | 83
Participants | 40 | 13

2. Secondary Outcome: Mean Change From Baseline in Corneal Endothelial Cell Density After Treatment With AG-920
Description: Endothelial cell count (and corneal morphology) will be summarized by continuous summaries
Time Frame: From Day 1 (treatment day) to 90 days following treatment
Measure: Mean (Standard Deviation); unit: cells/mm2
Arm/Group | AG-920 | Placebo
Number analyzed (Participants) | 13 | 3
cells/mm2 | -23.83 (92.18) | -44.33 (85.19)

ADVERSE EVENTS:
Time Frame: Adverse events were reported starting from the time of signing the informed consent until the end of the study assessment (follow up phone call at day 2-5 or day 90 for specular microscopy subjects).
Arm/Group | AG-920 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/83
Other Adverse Events (participants affected / at risk) | 38/166 | 10/83
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG-920 (N=166) | Placebo (N=83)
Instillation site pain (General disorders) | 38 (38) | 10 (10) — General disorders and administration site conditions - Instillation site pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigative site, the Principal Investigator, and any other investigators understand and agree that the Study is a multi-center clinical study and that a multicenter publication may be prepared and published by the Sponsor. The investigative site and its investigators will not, individually or together, present or publish any findings, data or results of the Study.

DOCUMENTS (2):
  • Study Protocol (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT05501860/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT05501860/SAP_001.pdf